CLINICAL TRIAL: NCT04265391
Title: Protein Supplementation of Snakehead Fish Cookies on Pregnant Women to Prevent Intrauterine Growth Restriction and Low Birth Weight in Sleman District, Yogyakarta Province, Indonesia: a Randomized Controlled Trial Study
Brief Title: Protein Supplementation of Snakehead Fish Cookies on Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Collaborators: Indonesia-MoH (Other Government)
Responsible Party: Principal Investigator, Eugenius Phyowai Ganap, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Snakehead fish cookies
Record Dates: First submitted 2020-02-04; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Pregnancy Related
Keywords: snakehead fish cookies; intrauterine fetal growth; low birth weight; randomized controlled trial; protein supplementation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Snakehead fish cookies (Experimental): Subjects who were given intervention of snakehead fish cookies during the study period
  Interventions: Dietary Supplement: cookies
- Standard cookies (Placebo Comparator): Subjects who were in control group and received standard cookies
  Interventions: Dietary Supplement: cookies

INTERVENTIONS:
Dietary Supplement: cookies — Either snakehead fish cookies or standard cookies were given to subjects 75g per day.

SUMMARY:
This study was randomized controlled trial study whose subjects were pregnant women in Sleman District, Yogyakarta, Indonesia. The aims of this study were to make snakehead fish cookies formula which can be well accepted by pregnant women and to observed its effect on fetal growth and birth weight and length. It was hypothesized that snakehead fish cookies could prevent intrauterine fetal growth (IUGR) and low birth weight (LBW).

Subjects on this study were randomly allocated into two groups which were treatment and control group. Subjects in treatment group were given snakehead fish cookies, while subject in control group received standard cookies. The intervention period lasted until subjects delivered their babies.

DETAILED DESCRIPTION:
Subjects were enrolled from Public Health Center (puskesmas) in Sleman District, Yogyakarta Province, Indonesia. Subjects were being explained about the study intervention and were given informed consent as an approval of joining this study. The intervention was given everyday as much as 75g cookies for several weeks period (until delivery). Examination on fetal growth was done every month for each subjects. Birth weight and length were collected after delivery from child health book record.

ELIGIBILITY:
Inclusion Criteria:

1. second and third trimester gestational age,
2. lower-class family with income under Sleman District minimum wage in 2019 (< 1,701,000 Rupiah),
3. pregnant women of under 25 years old, and
4. high school graduate or below

Exclusion Criteria:

1. suffering from anemia,
2. experiencing preeclampsia,
3. having multiple gestational, and
4. allergic to fish, eggs, and chocolate.

Max Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Estimated fetal weight (EFW) | change from baseline EFW after 1 month
  We measured EFW monthly using 2D ultrasonography (USG) for each subjects
Biparietal diameter (BPD) | change from baseline BPD after 1 month
  We measured BPD monthly using 2D ultrasonography (USG) for each subjects
Abdominal circumference (AC) | change from baseline AC after 1 month
  We measured AC monthly using 2D ultrasonography (USG) for each subjects
Femur length (FL) | change from baseline FL after 1 month
  We measured FL monthly using 2D ultrasonography (USG) for each subjects
Birth weight | immediately after the baby is born
  Birth weight of the baby
Birth length | immediately after the baby is born
  Birth length of the baby

CONTACTS AND LOCATIONS:
Overall Officials: Eugenius P Ganap, PhD, Principal Investigator — Gadjah Mada University
Locations (1):
- Public Health Center (Puskesmas) in the area of Sleman District, Sleman, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
This research was supported by Ministry of Health of Indonesia, and all data collected in this study were subject to Indonesian Ministry of Health rights.